CLINICAL TRIAL: NCT04474730
Title: Physical Activity Monitoring Among Bone Marrow Transplant Patients: An Apple Watch Feasibility Study
Brief Title: Physical Activity Monitoring Among BMT Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ming-Yuan Chih (Other)
Responsible Party: Sponsor-Investigator, Ming-Yuan Chih, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 51563
Record Dates: First submitted 2020-06-15; First posted 2020-07-17 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Bone Marrow Transplantation
Keywords: Bone Marrow Transplantation; Mobile Health; Symptom Management; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: In this study, we conduct a small randomized controlled trial to study the feasibility of an Apple Watch app developed to monitor bone marrow transplant patients' physical activities at their initial hospitalization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Watch Only (Active Comparator)
  Interventions: Other: Watch Only
- Watch+App (Experimental)
  Interventions: Device: BMT Physical Activity app

INTERVENTIONS:
Device: BMT Physical Activity app — This app sends reminders to patients, collect activity data from Apple Watch, and allow patients to submit symptoms.
  Arms: Watch+App
Other: Watch Only — A locked Apple Watch will be used to collect physical activity data from the Watch Only patients.
  Arms: Watch Only

SUMMARY:
This study aims to evaluate the feasibility of an apple watch-based application to promote physical activity among bone marrow transplant (BMT) patients.

DETAILED DESCRIPTION:
The research objective is to test the feasibility of using an Apple Watch-based system with the capacity to monitor BMT patients' physical activity and other patient reported outcomes at an ongoing basis within the inpatient BMT setting at the University of Kentucky Markey Cancer Center (UKMCC). The central hypothesis in this project is that the Apple Watch-based system designed based on user-centered design principles and the proposed study method will yield high feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Design Phase: Post 100 days BMT patients, family caregivers and providers
* Trial Phase: New BMT patients

Exclusion Criteria:

* under 18 years old;
* can't communicate, read or write in English;
* having any communicable infection or showing the signs of it, including coughing, fever, or rash;
* and incapable of completing the assigned research activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment | The day of recruitment
  Recruitment rate: the percentage of eligible patients who are enrolled
Feasibility - Study completion | From enrollment to 30 day post transplant or at hospital discharge
  Study completion rate - The percentage of enrolled patients who completed the study
Feasibility - Usability | 30 day post transplant or at hospital discharge
  A survey scale (User version - Mobile Application Rating Scale or uMARS) will be used to measure usability. uMARS scale score is calculated by averaging the likert scale answers, which range from 0 to 5. The uMARS score of 3.5 or higher is deemed to be acceptable usability.

SECONDARY OUTCOMES:
Physical Activity | 30 days post intervention or at hospital discharge
  Steps

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chih, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No